CLINICAL TRIAL: NCT06267144
Title: Dynamic Monitoring of MRD in Neoadjuvant Chemoimmunotherapy for Resectable Stage II-IIIB Non-small Cell Lung Cancer：An Observational Study
Brief Title: Detection of Minimal Residual Disease in Resectable Stage II-IIIB Non-small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 23K237-001
Record Dates: First submitted 2024-01-22; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer
Keywords: Neoadjuvant; Non Small Cell Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- immunotherapy and chemotherapy: Participants received two to three cycles of neoadjuvant chemoimmunotherapy before surgery. Adjuvant chemotherapy was also administered for 2-3 cycles after surgery. In addition, MRD was detected within 30 days before surgery, 1 week after surgery, 1 month ±7days after surgery, 6 months after surgery.
  Interventions: Drug: Sintilimab plus chemotherapy

INTERVENTIONS:
Drug: Sintilimab plus chemotherapy — Sintilimab: 200 mg via intravenous infusion on Day 1 of each 21-day cycle for 2-3 cycles in the neoadjuvant therapy and the maintenance therapy.
  Chemotherapy drugs: carboplatin/cisplatin+Pemetrexed/gemcitabine/albuminpaclitaxel.
  Carboplatin: AUC 5 via intravenous infusion, administered in 3-week (21 days) cycles for 2-3 cycles before and after surgery respectly.
  Cisplatin: 75 mg/m2 via intravenous infusion, administered in 3-week (21 days) cycles for 2-3 cycles before and after surgery respectly.
  Pemetrexed: 500mg/m2 via intravenous infusion, administered in 3-week (21 days) cycles for 2-3 cycles before and after surgery respectly.
  Gemcitabine:1.0g/m2 via intravenous infusion in day1 and day8, administered in 3-week (21 days) cycles for 2-3 cycles before and after surgery respectly. Albuminpaclitaxel: 260 mg/m2 via intravenous infusion, administered in 3-week (21 days) cycles for 2-3 cycles before and after surgery respectly.

SUMMARY:
Predicting relapse and overall survival in potentially resectable Stage IIIA-IIIB Non-small Cell Lung Cancer (NSCLC) patients remains challenging. It is now widely recognized that patients with detectable MRD have a worse prognosis than those with undetectable MRD. Therefore, investigators performed this prospective clinical trial to evaluate the predictive value of MRD with increased risk of relapse and improves prediction of outcome in potentially resectable Stage IIIA-IIIB NSCLC with neoadjuvant chemoimmunotherapy. In this study, investigators will pay more attention to the long-term follow-up time and dynamic monitoring of MRD. The predictive value of MRD with Disease-free survival (DFS) rate was observed as the primary endpoint. Besides that, the correlation of MRD with major pathologic response (MPR) rate, pathologic complete response (pCR) rate，event-free survival(EFS) rate and overall survival (OS) were observed as the second endpoints. Investigators hope it will provide a new insight for these potentially resectable Stage IIA-IIIB NSCLC with neoadjuvant chemoimmunotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 2.
* Have previously untreated and histological examination confirms resectable stage II-IIIA/IIIB non-small cell lung cancer (according to the 8th edition of the AJCC TNM staging criteria), and the pathological type of squamous cell carcinoma and non-squamous cell carcinoma needs to be distinguished, and EGFR, ALK, and ROS1 should be negative for non-squamous non-small cell lung cancer
* Adequate organ function and expected survival time ≥ 12 weeks;
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients.

Key Exclusion Criteria:

* Presence of mixed carcinoma component on histology.
* Patients with other active malignancies within 5 years prior to enrollment.
* Known active autoimmune diseases.
* Currently participate in an interventional clinical study treatment or have been treated with another drug or investigational device within 4 weeks prior to the first dose.
* Use of immunosuppressive agents within 14 days prior to the first dose of study treatment.
* Presence of other uncontrolled serious medical conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient initially diagnosed with resectable stage III-IIIA/IIIB non-small cell lung cancer t the First Hospital of Jilin University.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-17 (Estimated)

PRIMARY OUTCOMES:
Event free survival(EFS) | Six months after the surgery
  Defined as the time from randomization to the occurrence of any event, including disease progression, discontinuation of treatment for any reason, or death

SECONDARY OUTCOMES:
Overall Survival (OS) | Six months after the surgery
  Defined as the time from the first dose of study drug to death due to any cause.
Objective Response Rate (ORR) | Six months after the surgery
  Defined as the percentage of participants having complete response or partial response to protocol treatment. Objective response will be measured by RECIST 1.1.
Disease-Control Rate (DCR) | Six months after the surgery
  Defined as the proportion of patients with complete response, partial response, and stable disease.
Pathological complete response rate（PCR） | At the end of 2-3 cycles of neoadjuvant therapy (each cycle is 21 days)
  Defined as the absence of residual tumor cells (RVT) in the tumor bed in the pathological response assessment of postoperative specimens after neoadjuvant therapy (the criterion of most studies also includes the absence of tumor residue in the lymph nodes).
Major pathological response rate (MPR) | At the end of 2-3 cycles of neoadjuvant therapy (each cycle is 21 days)
  Defined as the proportion of residual surviving tumor cells in the tumor bed in the postoperative specimen is less than or equal to 10%.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital Of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No